CLINICAL TRIAL: NCT02365181
Title: A Randomized Controlled Non-inferiority Trial Between the Intra-articular Local Anesthetic Infiltration With Catheter and Interscalene Block With Catheter in Postoperative Analgesia After Shoulder Prosthesis
Brief Title: A Trial Between the Intra-articular Local Anesthetic Infiltration With Catheter and Interscalene Block With Catheter in Postoperative Analgesia After Shoulder Prosthesis
Acronym: LIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician responsible of clinical research, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APR092014
Record Dates: First submitted 2015-02-06; First posted 2015-02-18 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
Keywords: Shoulder arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IAL (Experimental): intra-articular local anesthetic infiltration with catheter
  Interventions: Procedure: intra-articular local anesthetic infiltration; Drug: Ropivacaine 2 %
- ISB (Active Comparator): interscalene block with catheter
  Interventions: Procedure: inter-scalene block; Drug: Ropivacaine 2 %

INTERVENTIONS:
Procedure: intra-articular local anesthetic infiltration — intra-articular local anesthetic infiltration with 20 ml of Ropivacaine 2 % and catheter
  Arms: IAL
Procedure: inter-scalene block — inter-scalene block with 20 ml of Ropivacaine 2 % and catheter
  Arms: ISB
Drug: Ropivacaine 2 % — 20 ml of Ropivacaine 2 %

SUMMARY:
The control of perioperative pain is necessary to avoid worst surgical suites after shoulder arthroplasty. Interscalene block (ISB) with or without catheter is the gold standard in postoperative analgesia after shoulder prosthesis but neurological or respiratory adverse events can occured . The intra-articular local (IAL) anesthetic infiltration with catheter is a simple procedure. Its efficacy was proved in knee and hip arthroplasty but not in shoulder arthroplasty. Our hypothesis was the IAL is as effective as ISB in early postoperative analgesia after shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder arthroplasty
* Osteoarthritis
* Consent

Exclusion Criteria:

* Previous surgery in the same shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean postoperative pain | during the 48 first hours

SECONDARY OUTCOMES:
Complications dues to anesthesia procedure | At 12 hours after surgery

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Polyclinique du Plateau, Bezons
  - Hospital Ambroise Paré Paris, Boulogne-Billancourt
  - Clinique Claude Bernard, Ermont
  - Clinique Jules Verne, Nantes
  - Institut Mutualiste Montsouris, Paris